CLINICAL TRIAL: NCT06503055
Title: Antibiotic Abuse Patterns: Medical Field And Population-Based Survey In Gharbia Governorate, Egypt
Brief Title: Antibiotic Abuse Patterns in Gharbia, Egypt
Status: Recruiting | Type: Observational
Sponsor: Rania Mamdouh Elkafoury (Other)
Responsible Party: Sponsor-Investigator, Rania Mamdouh Elkafoury, Sponsor-Investigator, Tanta University
Organization: Tanta University (Other)
Other Study IDs: 36264PR630/4/24
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Antibiotic Abuse
Keywords: Antibiotic abuse; Antibiotic resistance
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: The questionnaire will target a convenience sample of the general population in the Gharbia governorate.
  Interventions: Other: Questionnaire
- Healthcare professionals: The questionnaire will target a convenience sample of healthcare professionals in the Gharbia governorate including physicians with different specialties, pharmacists, medical students, and nursing staff.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire targeting a convenience sample of medical field professionals including physicians with different specialties, pharmacists, medical students, nursing staff, and the general population in Gharbia governorate (about 1000 subjects).
  The questionnaire will be written and digital in both Arabic and English versions. Moreover, an awareness campaign will be designed to educate the participants on appropriate antibiotic use principles.

SUMMARY:
Antimicrobial resistance (AMR) represents a serious problem described by the World Health Organization (WHO) as "a global public health concern". Research from around the globe indicates high rates of practices related to injudicious use of antibiotics as leftover antibiotics, antibiotic non-adherence, the pressure made by patients who request antibiotics from clinicians, unwarranted provision of antibiotics by physicians and pharmacists, antibiotic abuse and misuse in the form of overuse or underuse.

Moreover, many patients believe they have the right to self-prescribe an antibiotic or get one from friends and family. About 50% of antibiotic use is done improperly using the wrong agent, dose, or duration.

In Egypt, antibiotic misuse and overuse led to a high prevalence of multidrug-resistant (MDR) bacteria among the population.

The current work aims to assess the prevalence of antibiotic abuse among medical field professionals and the public and understand the factors leading to antibiotic misuse, thus evaluating awareness levels regarding antibiotic resistance.

DETAILED DESCRIPTION:
This scientific research will be done by a collaboration of both the Tropical Medicine Department and the Public Health Department, at Tanta University Hospital as a cross-sectional study using a digital and written questionnaire, this questionnaire will target medical field professionals and the public in Gharbia governorate.

Type of study:

Prospective, cross-sectional survey.

Duration of study:

The study will be carried out from May 2024 to August 2024 or until the target number is reached.

Target subjects:

The questionnaire will target a convenience sample of medical field professionals and the public in the Gharbia governorate including physicians with different specialties, pharmacists, medical students, nursing staff, and the general population (about 1000 subjects).

The questionnaire will be written and digital in both Arabic and English version. Moreover, an awareness campaign will be designed to educate the participants on appropriate antibiotic use principles.

Methodology:

After designing the questionnaire, it will be discussed with other experts in this field, where the validity and reliability will be assessed, and a pilot study will be done.

After informed consent, the subject will answer a designed questionnaire either written or digital. 2 phases will be done Phase 1: The questionnaire will be divided into 3 sectors Sector 1: Demographic data: questions about (age, sex, residence, educational level, occupation (subspeciality), workplace for all participants.

Sector 2: Socioeconomic level determination mainly for population :( Socio-economic data as the number of family members, rooms in the apartment, level of education, occupation, and cost per month).

Sector 3: the main work includes questions for the population: (behavior of seeking medical advice, the last use of antibiotic, type and duration, adherence to the prescribed regimen, who prescribed and why, side effects, if there are any laboratory investigations done to determine the correct antimicrobial use, duration between 2 consequent antibiotic use, number of antibiotic used in the last time and how many times of antibiotic use in the last six months).

For prescriber :( most type of antibiotic used in the last six months, how many times antibiotic was prescribed, patient criteria for whom antibiotic prescribed, any lab done to determine the propitiate antibiotic, durations of antibiotic prescription, perception of patients to the prescribed antibiotic, patients stress in demanding antibiotic prescription, the outcome of this prescription, duration between 2 consequent prescriptions in the same patient and use of more than one combination in the same patient within the same time) Phase 2: An awareness campaign will be designed to educate the participants on appropriate antibiotic use principles.

Ethical considerations:

A written or digital informed consent form authorizing the collection of this data will be signed by all subjects The study will be approved by the Ethical Committee of the Faculty of Medicine at Tanta University.

The risks to the participants and measures needed to minimize these risks:

* The privacy of the data of the patients will be maintained(the procedure will be discussed later in this protocol
* Any unexpected risks that appear during research will be cleared to the subjects and the ethical committee on time

Adequate provisions to maintain the privacy of participants and confidentially of data are as follows:

* A code number for each patient will be used, and symbols for the name and address will be kept in a special file.
* The patients' names will be hidden when we use the research
* The research results will be used only for scientific aims and not for other aims.

ELIGIBILITY:
Inclusion Criteria:

* All medical field professionals and students with any specialty can participate in the survey
* Population more than 18 years old
* Parents of children less than 18 years old.

Exclusion Criteria:

* Participants outside the Gharbia governorate.
* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire will target a convenience sample of medical field professionals and the public in the Gharbia governorate including physicians with different specialties, pharmacists, medical students, nursing staff, and the general population (about 1000 subjects).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
prevalence of antibiotic abuse | till August 2024
  using a questionnaire to assess prevalence of antibiotic abuse among both medical field professionals and the public.

SECONDARY OUTCOMES:
factors leading to antibiotic misuse | till August 2024
  using a questionnaire to understand the factors leading to antibiotic misuse.
awareness of antibiotic resistance | till August 2024
  using a questionnaire to evaluate awareness levels about antibiotic use and antibiotic resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Tanta University Hospitals, Tanta, Gharbyea, Egypt